CLINICAL TRIAL: NCT07054814
Title: Effect Of Games Based Virtual Reality On Promoting Early Functional Recovery After Foot Tendon Repair
Acronym: VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Araby Osman Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mohamed-0055846
Record Dates: First submitted 2025-06-28; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Virtual Reality; Achilles Tendon Repairs/Reconstructions
Keywords: Achilles tendon repair

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (participant )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gemes based virtual reality (Experimental): This group includes 30 patients who will receive game based virtual reality exercise using samsung Gear VR plus accelerate functional rehab programe physical therapy 3 times per week for 30 minutes for 12 weeks starting once patient able to do partial or complete weight bearing around (4-6 weeks post operative).
  Interventions: Device: samsung gear VR google; Other: Traditional theraapy
- accelerated functional rehab protocol (Active Comparator): This group includes 30 patients who will receive accelerated functional rehab programe only for 3 sessions per week .
  Interventions: Other: Traditional theraapy

INTERVENTIONS:
Device: samsung gear VR google — do some of games based VR exercise Headmaster 3.0 Dream Match Tennis Beat Saber (PSVR) Knockout League Hoops Richie's Plank Experience Pong It VR Egg Time VR Sparc VR plus accelerated functional rehab protocol
  General Principles:
  Goal: Promote tendon healing while minimizing stiffness, muscle atrophy, and encouraging a faster return to full function.
  Approach: Early controlled mobilization, gradual loading based on patient tolerance (without excessive pain or swelling).
  Important: Supervised by an orthopedic surgeon and a physical therapist. Device: Start with a walker boot or splint keeping the ankle plantarflexed.
  Phases of Rehabilitation:
  Other Names: traditional protocol of accelerated functional rehab
  Arms: gemes based virtual reality
Other: Traditional theraapy — General Principles: accelerated functional rehab protocol Goal: Promote tendon healing while minimizing stiffness, muscle atrophy, and encouraging a faster return to full function.
  Approach: Early controlled mobilization, gradual loading based on patient tolerance (without excessive pain or swelling).
  Important: Supervised by an orthopedic surgeon and a physical therapist. Device: Start with a walker boot or splint keeping the ankle plantarflexed.
  Phases of Rehabilitation:

SUMMARY:
The purpose of this study is to investigate the effectiveness of integrating game based virtual reality on muscle strength ,balance , range of motion ,functional mobility after foot tendon repair and to compare it with standard rehabilitation methods.

DETAILED DESCRIPTION:
This research is significant for several reasons:

1. Clinical Impact: It seeks to provide evidence-based insights into the effectiveness of VR in enhancing rehabilitation outcomes, potentially reducing recovery times and improving functional independence for patients.
2. Technological Advancement: By integrating cutting-edge technologies into rehabilitation, this study contributes to the evolution of personalized and immersive therapeutic approaches.
3. Patient-Centered Care: The findings may lead to more engaging and accessible rehabilitation options, improving adherence and satisfaction among patients.
4. Healthcare Efficiency: Successful integration of these technologies could reduce the burden on healthcare systems by shortening rehabilitation durations and decreasing the need for extensive manual interventions.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 26 years. Patients undergoing or who have undergone unilateral achilles tendon surgical repair .

4-6 weeks post operative ,partial to full weight bearing Patients willing to participate in rehabilitation protocol.

-

Exclusion Criteria:

* o Patients with severe diseases or impaired control of gait patterns.

  * Patients with high scores in anxiety or stress tests, indicating significant psychological distress.
  * Patients who report fatigue or are medically unstable.
  * Patients who have any other orthopedic or neurological problems .
  * Patients who have renal, cardiac,hepatic edema
  * Patients who have gout,plantar fasciitis,fracture dislocation or any types of foot ulcer.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Balance | At base line and 6 weeks
  Biodex balance system for balance assessment

SECONDARY OUTCOMES:
Symptom relief | At base line and at 6 and 12 week
  Visual analogue scale
Range of motion | At baseline and at 6 weeks and 12 weeks
  Goniometer
Functional ability | At base line and at 6 weeks and at 12 weeks
  6 minute walk test
Symmetry | At base line and week 6 and wee12
  Limb symmetry index
Muscle strength | At baseline and week 6 and 12
  Hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AR Osman, MSC, Principal Investigator — Police hospital ,cairo ,egypt
Locations (1):
- Police Hospital Ministry of Interior, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No